CLINICAL TRIAL: NCT03796442
Title: Early and 1-year Hemodynamic Performance and Clinical Outcomes After Aortic Valve Replacement Using Two Pericardial Bioprostheses: A Multicenter Randomized Controlled Trial
Brief Title: Comparison of Two Pericardial Bioprostheses in AVR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Ho Young Hwang, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D-1812-024-991
Record Dates: First submitted 2019-01-01; First posted 2019-01-08 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Aortic Valve Disease
Keywords: aortic valve replacement; bioprosthesis
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- AVALUS group (Experimental): patients who will undergo aortic valve replacement with Avalus bioprosthesis
  Interventions: Device: AVR with AVALUS
- CEPME group (Active Comparator): patients who will undergo aortic valve replacement with Carpentier-Edwards Perimount Magna Ease bioprosthesis
  Interventions: Device: AVR with CEPME

INTERVENTIONS:
Device: AVR with AVALUS — aortic valve replacement with AVALUS bioprosthesis
  Arms: AVALUS group
Device: AVR with CEPME — aortic valve replacement with Carpentier-Edwards Perimount Magna Ease bioprosthesis
  Arms: CEPME group

SUMMARY:
The purpose of the study is to compare early and 1-year hemodynamic performance and clinical outcomes after aortic valve replacement using two pericardial bioprosthesis, Avalus and Carpentier Edwards Perimount Magna Ease.

DETAILED DESCRIPTION:
This trial was designed as a multicenter randomized, controlled trial to recruit 386 patients who undergo aortic valve replacement with pericardial bioprosthesis. Patients were randomized by use of a randomization table. Bioprosthesis was chosen between Avalus or Carpentier Edwards Perimount Magna Ease according to the randomization result. The primary end point is postoperative 1-year transvalvular mean pressure gradient. The secondary end points are postoperative 1-year effective orifice area, operative mortality, operative morbidities, 1-year overall survival, 1-year freedom from cardiac death and 1-year freedom from valve-related events.

ELIGIBILITY:
Inclusion Criteria:

* patients who are going to undergo aortic valve replacement with bioprosthesis

Exclusion Criteria:

* heart failure with severe LV dysfunction (LV EF <30%)
* active infective endocarditis
* with other critical cardiovascular disease (e.g. acute aortic dissection)
* with other critical comorbities by which the expected life span is less than 1 year
* inadequate participant by the researcher's discretion

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2021-05-13 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ho Young Hwang, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared because it is not allowed by our institutional IRB.

REFERENCES:
- [Derived] Sohn SH, Kang Y, Kim JS, Choi JW, Lee JH, Kim JS, Lim C, Hwang HY. A Controlled Trial Comparing One-Year Hemodynamics of Two Bovine Pericardial Valves. Thorac Cardiovasc Surg. 2025 Mar;73(2):132-140. doi: 10.1055/a-2199-2087. Epub 2023 Oct 26. PMID 37884030
- [Derived] Sohn SH, Kim JS, Choi JW, Lee JH, Kim JS, Lim C, Hwang HY. Preliminary Report from a Randomized Controlled Trial Comparing Two Bovine Pericardial Valves. Thorac Cardiovasc Surg. 2023 Dec;71(8):648-655. doi: 10.1055/s-0042-1753494. Epub 2022 Aug 2. PMID 35917824

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AVALUS Group | CEPME Group
Started | 70 | 70
Completed | 66 | 63
Not Completed | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AVALUS Group | CEPME Group | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.4 (5.5) | 74.3 (6.9) | 72.8 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 33 | 69
  Male | 34 | 37 | 71
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 70 | 70 | 140
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 70 | 70 | 140
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 24.8 (3.4) | 24.4 (2.8) | 24.6 (3.1)
Body surface area [Mean (Standard Deviation); unit: m^2] | 1.64 (0.18) | 1.65 (0.15) | 1.65 (0.16)
Diabetes mellitus [Count of Participants; unit: Participants] | 24 | 24 | 48
Hypertension [Count of Participants; unit: Participants] | 52 | 47 | 99
Dyslipidemia [Count of Participants; unit: Participants] | 42 | 31 | 73
Chronic obstructive pulmonary disease [Count of Participants; unit: Participants] | 4 | 9 | 13
Stroke [Count of Participants; unit: Participants] | 7 | 7 | 14
Chronic kidney disease [Count of Participants; unit: Participants] | 8 | 18 | 26
Peripheral vascular disease [Count of Participants; unit: Participants] | 1 | 2 | 3
Atrial fibrillation [Count of Participants; unit: Participants] | 8 | 7 | 15
Reoperation [Count of Participants; unit: Participants] | 1 | 1 | 2
EuroSCORE II [Mean (Standard Deviation); unit: units on a scale] — The EuroSCORE II (European System for Cardiac Operative Risk Evaluation) is a prognostic scoring system developed in Europe for patients undergoing cardiac surgery. It calculates the risk of in-hospital mortality after major cardiac surgery. The scale ranges from 0 to 100. Higher value of the EuroSCORE II represents that the patient is predicted to have a worse outcome.
  units on a scale | 1.87 (1.41) | 2.11 (1.67) | 1.99 (1.54)

OUTCOME MEASURES:

1. Primary Outcome: Transvalvular Mean Pressure Gradient (mPG)
Description: transvalvular mean pressure gradient measured by trans-thoracic echocardiography
Time Frame: at postoperative 1 year
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AVALUS Group | CEPME Group
Number analyzed (Participants) | 66 | 63
mmHg | 14.1 (4.3) | 13.9 (5.1)
Statistical Analysis 1: Comparison: AVALUS Group vs CEPME Group; The null hypothesis was that the AvalusTM was inferior to the CEPME based on the AVMPG at 1-year echocardiographic follow-up, with a non-inferiority margin of 3mmHg. The result for the primary endpoint was presented with 97.5% one-sided confidence interval for mean difference between groups. The non-inferiority test was performed using a t-test which compared mean difference between groups with the non-inferiority margin under the one-sided significance level of 0.025; Test type: Non-Inferiority — The study was designed to have 80% power to detect 1-year AVMPG of 12.6±4.3mmHg for the study prosthesis and 11.9±4.3mmHg for the control prosthesis, with a 1-sided type I error of 2.5% and a noninferiority margin of 3mmHg. The noninferiority margin was determined by the values of 15mmHg for AVMPG of clinically significant aortic stenosis and 12mmHg for AVMPG of the control prosthesis; p = 0.0004, t-test, 1 sided

2. Secondary Outcome: Effective Orifice Area (EOA)
Description: effective orifice area measured by trans-thoracic echocardiography
Time Frame: at postoperative 1 year
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | AVALUS Group | CEPME Group
Number analyzed (Participants) | 66 | 63
cm2 | 1.48 (0.39) | 1.53 (0.38)

3. Secondary Outcome: Number of Participants With Op Mortality
Description: any death within 30 days after surgery or during the same hospital admission
Time Frame: at postoperative 30 days or at the time of discharge
Measure: Count of Participants; unit: Participants
Arm/Group | AVALUS Group | CEPME Group
Number analyzed (Participants) | 70 | 70
Participants | 0 | 0

4. Secondary Outcome: Number of Participants With Op Morbidities
Description: low cardiac output syndrome, bleeding reoperation, perioperative myocardial infarction, stroke, acute kidney injury, respiratory complication, new onset atrial fibrillation, mediastinitis, surgical wound infection
Time Frame: at postoperative 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | AVALUS Group | CEPME Group
Number analyzed (Participants) | 70 | 70
Participants
  Postoperative atrial fibrillation | 21 | 24
  Respiratory complication | 6 | 7
  Acute kidney injury | 4 | 2
  Stroke | 2 | 2
  Low cardiac output | 2 | 1
  Complete atrioventricular block | 2 | 0
  Bleeding reoperation | 1 | 1
  Mediastinitis | 0 | 0
  Infective endocarditis | 0 | 0
  No complication | 32 | 33

5. Secondary Outcome: Number of Participants With All-cause Mortality
Description: patients who died from any cause
Time Frame: at postoperative 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | AVALUS Group | CEPME Group
Number analyzed (Participants) | 70 | 70
Participants | 1 | 6

6. Secondary Outcome: Number of Participants With Cardiac Death
Description: Any death related to cardiac events, including sudden death during follow-up
Time Frame: at postoperative 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | AVALUS Group | CEPME Group
Number analyzed (Participants) | 70 | 70
Participants | 1 | 2

7. Secondary Outcome: Number of Participants With Aortic Valve-related Events
Description: valve-related mortality, thromboembolism, bleeding, endocarditis, reoperation
Time Frame: at postoperative 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | AVALUS Group | CEPME Group
Number analyzed (Participants) | 70 | 70
Participants | 5 | 6

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | AVALUS Group | CEPME Group
All-Cause Mortality (participants affected / at risk) | 1/70 | 6/70
Serious Adverse Events (participants affected / at risk) | 5/70 | 6/70
Other Adverse Events (participants affected / at risk) | 0/70 | 0/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AVALUS Group (N=70) | CEPME Group (N=70)
cardiac deaths (Cardiac disorders) | 1 | 2
nonstructural valve dysfunction (Cardiac disorders) | 1 | 3
thromboembolism (Cardiac disorders) | 0 | 2
bleeding event (Cardiac disorders) | 1 | 0
prosthetic valve endocarditis (Cardiac disorders) | 2 | 1
permanent pacemaker implantation (Cardiac disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-12-28): https://cdn.clinicaltrials.gov/large-docs/42/NCT03796442/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-28): https://cdn.clinicaltrials.gov/large-docs/42/NCT03796442/SAP_001.pdf